CLINICAL TRIAL: NCT06125535
Title: Biomolecular Phenotyping of Lung Transplant Recipients: a Prospective Observational Study
Brief Title: Biomolecular Phenotyping of Lung Transplant Recipients
Acronym: LUTX_phenotype
Status: Completed | Type: Observational
Sponsor: Policlinico Hospital (Other)
Collaborators: University of Milan (Other)
Responsible Party: Principal Investigator, Giacomo Grasselli, Prof, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: LUTX_phenotype
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Lung Transplant Failure
Keywords: lung transplant; primary graft dysfunction; prospective observational study; biomarkers
MeSH Terms: conditions — Primary Graft Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples collected at <6 hours and 36 hours from graft reperfusion. Fresh-frozes. Biobanked at -80°c
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypoinflammatory: By means of latent class analysis, a sub-phenotype of LUTX recipients with down-regulated inflammatory biomarkers
  Interventions: Diagnostic Test: Sub-phenotyping by biomarkers concentration
- Hyperinflammatory: By means of latent class analysis, a sub-phenotype of LUTX recipients with up-regulated inflammatory biomarkers
  Interventions: Diagnostic Test: Sub-phenotyping by biomarkers concentration

INTERVENTIONS:
Diagnostic Test: Sub-phenotyping by biomarkers concentration — Plasma will be collected at ICU admission (i.e., < 6 hours from graft reperfusion), centrifuged (1500G for 15 min), frozen at -80°c, and then centralized at the Institutional laboratory. The following biomarkers will be assessed: Interleukin-1β, Interleukin-2, Interleukin-6, Interferon-γ, Tumor Necrosis Factor-alpha (TNF-α), chemokine (C-C motif) ligand-2 (CCL-2), Interleukin-15 (IL-15), Ferritin, and D-dimer, by a point-of-care biochip-array device (RANDOX, Multistat)

SUMMARY:
Primary graft dysfunction (PGD) is a common problem after a lung transplant. It's a sudden lung injury that affects around 30% of patients within 72 hours of getting a new lung. PGD can vary in severity, from mild issues seen on X-rays to severe lung problems, and it can also affect other parts of the body, like the heart and kidneys.

The investigators believe that using precision medicine can identify different groups of patients with varying levels of inflammation and provide them with treatments tailored to their specific conditions. This approach has been successful in treating other serious conditions like acute respiratory distress syndrome (ARDS). Currently, researchers haven't classified lung transplant patients in this way, and there's limited information on early blood markers for PGD.

In an upcoming study, the investigators aim to group lung transplant patients based on their blood markers related to inflammation, blood clotting, and blood vessel problems. The investigators also want to see if these groups are linked to their overall outcomes, especially when it comes to PGD.

DETAILED DESCRIPTION:
Primary graft dysfunction (PGD) is the most common complication after lung transplant (LUTX). PGD is an acute form of lung injury with an incidence of 30%, defined upon alteration of oxygenation and radiographic criteria occurring <72 hours after graft reperfusion.

The PGD definition does not consider the heterogeneity of clinical manifestations of ischemia-reperfusion (I/R) injury. First, PGD severity may vary from mild radiographic signs to life-threatening lung injury. Second, duration may differ: most patients manifest transient hypoxia, but a minority have persistent respiratory failure. Finally, PGD is associated with hemodynamic and renal failure, suggesting that it might be considered a heterogeneous syndrome characterized by multisystemic widespread endothelial barrier damage and inflammation activation due to I/R injury rather than an alteration of the sole lung function.

Following the new paradigm of precision medicine, the investigators hypothesize that predictive enrichment may allow for detecting different - and potentially treatable - traits (i.e., hypo vs. hyperinflammatory) of PGD and applying targeted treatments to sub-cohorts. As for other critical illnesses (i.e., acute respiratory distress syndrome - ARDS, sepsis), the investigators envision the possibility of carrying out biological subtyping of LUTX patients to select the patients with the lowest chance of harm for treatment. In the similar -but not equivalent- context of ARDS, it has been proven that treatments (e.g., positive end-expiratory pressure, fluid management, simvastatin) that disappointingly failed to benefit the overall patients' population provided benefit in specific patients' subcohorts. Biological phenotyping of LUTX recipients has never been carried out, and literature is ample but sparse regarding early PGD plasmatic biomarkers.

With this prospective observational study, the investigators aim to assess: 1/ whether LUTX recipients can be clustered based on early plasma concentration of biomarkers of inflammation, coagulation, and endothelial activation, and 2/ whether these clusters could be associated with clinical outcomes (and specifically PGD).

ELIGIBILITY:
Inclusion Criteria:

* undergone double LUTX
* age > 18 years old

Exclusion Criteria:

* single LUTX
* re-transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the consecutive adult patients have undergone primary double LUTX at the promoting institution.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Primary Graft Dysfunction | <= 72 hours from graft reperfusion
  PGD incidence, defined and graded following the most recent ISHLT society guidelines, as hypoxia (i.e., PaO2/FiO2 < 300 mmHg) with bilateral lung infiltrates.

SECONDARY OUTCOMES:
28-days organ support free-days | 28 days from ICU admission
  Number of days at 28 days from ICU admission free from: - extracorporeal membrane oxygenation; - mechanical ventilation; - renal replacement therapy; - vasoactive support.

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Grasselli, Porf, Study Director — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico; Vittorio Scaravilli, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca'Granda - Ospedale Maggiore Policlinico, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual anonymized data will be available from the promoting center after a reasonable request
Supporting Information: Analytic Code
Time Frame: Any timeframe
Access Criteria: Request to the PI